CLINICAL TRIAL: NCT03531099
Title: Phase 3, Multicenter, Randomized Study, Evaluating the Efficacy and Tolerability of Focused HIFU Therapy Compared to Active Surveillance in Patients With Significant Low Risk Prostate Cancer
Brief Title: Phase 3, Multicenter, Randomized Study, Evaluating the Efficacy and Tolerability of Focused HIFU (High Intensity Focused Ultrasound) Therapy Compared to Active Surveillance in Patients With Significant Low Risk Prostate Cancer
Acronym: HIFUSA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL18_0203; 2018-A01024-51 (Other: ID-RCB)
Record Dates: First submitted 2018-05-09; First posted 2018-05-21 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; HIFU focal; adverse effect; low risk
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Therapeutics; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFU treatment (Experimental): 65 patients will receive the immediate treatment with focal HIFU in order to destroy the cancer without causing side effects. HIFU treatment will be conducted with the Focal One® device. The treatment area will be defined using MRI data and 3D biopsies. A safety distance of at least 9 mm will be defined around the tumor. An intraoperative contrast echocardiographic control will be performed to evaluate the necrotic area. If necessary, additional HIFU lesions will be performed during the same session. In case of residual tumor demonstrated during control biopsies, additional treatment of this tumor with focal HIFU may be proposed.
  Patients randomized in this arm will also have PSA dosage, MRI exam, questionnaires and prostatic biopsies during their follow up.
  Interventions: Procedure: treatment with focal HIFU; Biological: PSA dosage; Device: MRI; Other: Questionnaires; Procedure: Prostatic biopsies
- Active surveillance (Active Comparator): 65 patients will be randomized to active surveillance and will have exactly the same follow-up as treated patients excepting the HIFU treatment.
  Active surveillance is a therapeutic option that shifts the eventual moment of curative treatment while remaining within a window of curability of the disease.
  Patients randomized in this arm will also have PSA dosage, MRI exam, questionnaires and prostatic biopsies during their follow up.
  Interventions: Biological: PSA dosage; Device: MRI; Other: Questionnaires; Procedure: Prostatic biopsies

INTERVENTIONS:
Procedure: treatment with focal HIFU — HIFU treatment will be conducted with the Focal One® device. The treatment area will be defined using MRI data and 3D biopsies. A safety distance of at least 9 mm will be defined around the tumor. An intraoperative contrast echocardiographic control will be performed to evaluate the necrotic area. If necessary, additional HIFU lesions will be performed during the same session. In case of residual tumor demonstrated during control biopsies, additional treatment of this tumor with focal HIFU may be proposed.
  Arms: HIFU treatment
Biological: PSA dosage — PSA dosage will be regularly performed during patient follow up thanks to blood sampling.
Device: MRI — MRI exam will be regularly performed during patient follow up.
Other: Questionnaires — Patients will have to complete five questionnaires during their follow up : QLQ-C30 (Quality of Life questionnaire), EPIC-26 (The Expanded Prostate Cancer Index Composite), IPSS (International Prostate Score Symptom), IIEF-5 (The International Index of Erectile Function), STAI-YB (State-Trait Anxiety Inventory)
Procedure: Prostatic biopsies — Prostatic biopsies will be regularly performed during patient follow up.

SUMMARY:
The percentage of malignant prostate tumors detected very early is constantly increasing and the number of well differentiated tumors, with small volume and low risk of progression increases. When a tumor of this type is identified, radical prostatectomy remains the reference treatment, but this treatment is not without side effects. Active surveillance is a strategy which aims at detecting an early development of the cancerous disease in order to propose curative treatment in a timely manner and thus improve specific survival. Patients are therefore re-evaluated each year by rectal examination, PSA (Prostate-Specific Antigen) assay. Active surveillance remains difficult to manage psychologically for both the patient and the practitioner, because of the lack of treatment on the one hand and a rate of non-curable cancers close to 50% when signs of progression trigger a radical treatment.

The aim of the focal treatment HIFU (High Intensity Focused Ultrasound) is to destroy the cancer without causing side effects in contrast to radical treatments. It is in this sense that it is positioned both as an alternative to radical surgery and as an alternative to active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Patient having been clearly informed of the study and having accepted, with sufficient reflection time, to participate by signing the informed consent form of the study.
* Age between 50 and 80 years with a life expectancy of more than 5 years. Patients between the ages of 75 and 80 will need to have G8 score > 14.
* Initial diagnosis of localized prostate cancer (T1c or T2a) with the following characteristics:

  * Only one Target tumor on MRI on a maximum of 2 contigous sextants. Case allowed:

    * If more than one target tumor on MRI, only one of them must be confirmed by targeted prostate biopsies.
    * If no target tumor on MRI, only 2 contigous sextants must be positive on prostate biopsies
  * A maximum tumor length> 3 mm or at least 3 positive biopsies on all biopsies performed (randomized biopsies and/or MRI/Ultrasound Fusion-Guided Prostate Biopsy).
  * Gleason 6 score (risk group 1 of the D'Amico classification).
  * Tumor positioned so that a safety distance of at least 9 mm from external sphincter can be defined during HIFU-FOCAL treatment in prostate tissue around the target.
* PSA ≤ 15ng / ml.
* Patient affiliated with health insurance or beneficiary of an equivalent plan.

Exclusion Criteria:

* Contraindications to treatment with HIFU-F:

  * Tumor not accessible.
  * Multiple intra prostatic calcifications inducing, on ultrasound, a shadow cone in the prostate preventing the penetration of ultrasound and thus the realization of the treatment.
  * History of pelvic irradiation
  * Presence of an implant (stent, catheter) located less than 1 cm from the treatment area.
  * Fistula of the urinary tract or rectum.
  * Anal or rectal fibrosis, anal or rectal stenosis or other abnormalities making it difficult to insert the Focal One® probe.
  * Anatomical abnormality of the rectum or rectal mucosa.
  * Patient with artificial sphincter, penile prosthesis or intra prostatic implant, eg stent.
  * History of intestinal inflammatory pathology.
  * Uro-genital infection in progress (the infection to be treated before HIFU treatment).
  * Anterior surgery at the level of the anus or rectum making the introduction of the probe impossible.
  * Allergy to latex.
  * Thickness of the rectal wall> 10mm.
* TURP indication. Bladder neck incision is allowed .
* Patient with a medical contraindication to Sonovue® injection.
* Patient with a medical contraindication on MRI.
* Patient already treated for prostate cancer (hormone therapy, radiotherapy, surgery).
* History of uncontrolled cancer and / or treated for less than 5 years (with the exception of basal cell skin cancer).
* History of sclerosis of the bladder neck or urethral stenosis.
* Patient with a several bleeding risk according to medical advice (patient with oral anticoagulant therapy must receive an alternative therapy if randomized in HIFU-F arm).
* Patients with unstable neurological pathology.
* Patient who has been treated for a therapeutic trial within 30 days of enrollment or who wishes to participate in an ongoing study that may interfere with this study.
* Legal person protected by law.
* Patient not able to understand the objectives of the study or refusing to comply with postoperative instructions.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2025-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
patient proportion who needed to seek radical treatment | 48 month
  The primary endpoint is the comparison between the 2 groups of the proportion of patient converting to a radical treatment at 48 months of follow-up. Conversion to a radical treatment is define as a medical decision based on the following criteria:
  * An increase in Gleason score to a score 7 (3 + 4) with bilateral involvement (Gleason 6 or 7).
  * An increase in the Gleason score to a score 7 (3 + 4) with tumor whose location is not compatible with a focal treatment (impossibility to apply safety margins of 9mm).
  * An increase in Gleason score to a score of 7 (4 + 3) or higher.
  * Risk of lymph node invasion> 5% (calculated with the MSKCC nomogram)
  * An extension of the tumor beyond the prostatic capsule (MRI and / or biopsies).
  * Appearance of pelvic ganglion metastases.

SECONDARY OUTCOMES:
proportion of patients needing additional treatment | 24 months
  The objective is to compare between the 2 groups the proportion of patients needing additional treatment (focal or radical) at 24 months. This includes patients who wish or require radical treatment (prostatectomy, radiotherapy), total focal treatment, focal treatment for patients in the active surveillance group or additional treatment for patients in the treatment group.
proportion of patients needing additional treatment | 48 months
  The objective is to compare between the 2 groups the proportion of patients needing additional treatment (focal or radical) at 48 months. This includes patients who wish or require radical treatment (prostatectomy, radiotherapy), total focal treatment, focal treatment for patients in the active surveillance group or additional treatment for patients in the treatment group.
rate of positive biopsies | 24 months
  The rate of positive biopsies in the untreated lobe and treated lobe evaluated and will be used to evaluate the oncological evolution at 24 months.
rate of positive biopsies | 48 months
  The rate of positive biopsies in the untreated lobe and treated lobe will be measured and will be used to evaluate the oncological evolution at 48 months.
clinically significant cancer rate | 24 months
  The clinically significant cancer rate (Gleason 7 or invasion of more than 3 biopsies or invasion> 3 mm regardless of Gleason) in the untreated lobe and the treated lobe will be measured and will be used to evaluate the oncological evolution at 24 months.
clinically significant cancer rate | 48 months
  The clinically significant cancer rate (Gleason 7 or invasion of more than 3 biopsies or invasion> 3 mm regardless of Gleason) in the untreated lobe and the treated lobe will be measured and will be used to evaluate the oncological evolution at 48 months.
Gleason score | 24 months
  Evolution of the Gleason score (appearance of Gleason ≥7) will be measured and will be used to evaluate the oncological evolution at 24 months.
Gleason score | 48 months
  Evolution of the Gleason score (appearance of Gleason ≥7) will be measured and will be used to evaluate the oncological evolution at 48 months.
Appearance of another cancerous focus in the other half of the prostate | 24 months
  Appearance of another cancerous focus in the other half of the prostate will be supervised and will be used to evaluate the oncological evolution at 24 months.
Appearance of another cancerous focus in the other half of the prostate | 48 months
  Appearance of another cancerous focus in the other half of the prostate will be supervised and will be used to evaluate the oncological evolution at 48 months.
Appearance of metastases | 24 months
  Appearance of metastases (lymph node or bone) will be supervised and will be used to evaluate the oncological evolution at 24 months.
Appearance of metastases | 48 months
  Appearance of metastases (lymph node or bone) will be supervised and will be used to evaluate the oncological evolution at 48 months.
Appearance of an extra capsular extension | 24 months
  Appearance of an extra capsular extension will be supervised and will be used to evaluate the oncological evolution at 24 months.
Appearance of an extra capsular extension | 48 months
  Appearance of an extra capsular extension will be supervised and will be used to evaluate the oncological evolution at 48 months.
Overall survival | 48 months
  Overall survival at 48 months will be measured from the date of inclusion to the date of death, all causes of death combined or the date of last new or point date to 48 months.
Prostate cancer specific survival | 48 months
  Prostate cancer specific survival at 48 months will be measured from the date of inclusion to the date of death related to prostate cancer or the date of last new or point date to 48 months
Recurrence free survival | 48 months
  Prostate cancer specific survival at 48 months will be measured from the date of inclusion to the date of first metastasis , or the date of last new or point date to 48 months
Proportion of serious adverse effect | 48 months
  comparison between the 2 groups of the proportion of serious adverse effect at 48 months
Quality of life score | over the 48 months
  quality of life will be compared between the two groups and assessed using the QLQC30 questionnaire
EPIC-26 score | over the 48 months
  urinary function will be compared between the two groups and assessed using the EPIC-26 questionnaire.
IPSS score | over the 48 months
  urinary function will be compared between the two groups and assessed using the IPSS questionnaire.
IIEF-5 score | over the 48 months
  Sexual function will be compared between the two groups and assessed using the IIEF-5 questionnaire
STAi-YB score | Over the 48 months
  Anxiety will be compared between the two groups and assessed using the STAi-YB questionnaire

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Polyclinique du parc Rambot, Aix-en-Provence
  - Clinique Saint-Vincent, Besançon
  - Service d'Urologie, Clinique Tivoli Ducos, Bordeaux
  - Groupe Hospitalier Pellegrin - CHU, Bordeaux
  - Service d'Urologie, CHU de Guebwiller Colmar, Colmar
  - Service d'Urologie CHRU de Lille, Hôpital HURIEZ, Lille
  - Service d'Urologie Générale de Santé - Hôpital Privé La Louvière, Lille
  - Service d'Urologie et Chirurgie de la Transplantation, Hôpital Edouard Herriot,, Lyon
  - Service d'urologie Assistance Publique - Hôpitaux de Marseille - Hôpital Marseille Nord, Marseille
  - Département d'Urologie, Institut Montsouris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Clinique Urologique Nantes Atlantis, Saint-Herblain
  - Service d'Urologie, Hôpital Foch, Suresnes
  - CHU de Toulouse - Hôpital de Rangueil, Toulouse